CLINICAL TRIAL: NCT06106022
Title: A Phase 1, Randomized, Parallel-group, Open-label, Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Vonoprazan (10 or 20 mg Once Daily) in Children Aged ≥ 6 to < 12 Years Who Have Symptomatic Gastroesophageal Reflux Disease
Brief Title: A Study to Evaluate Vonoprazan in Children Who Have Symptomatic Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VPED-103; 2022-003228-42 (EudraCT Number)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastrology; Vonoprazan; Gastroesophageal Reflux Disease; Children; GERD; Pharmacokinetics
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vonoprazan 10mg (Experimental): Participants will receive vonoprazan 10mg QD for 14 days.
  Interventions: Drug: Vonoprazan
- Vonoprazan 20mg (Experimental): Participants will receive vonoprazan 20mg QD for 14 days.
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Administered orally

SUMMARY:
The aim of this study is to evaluate the pharmacokinetic (PK) profile of vonoprazan (10 or 20 mg once daily [QD]) in children ≥ 6 to < 12 years of age who have symptomatic Gastroesophageal Reflux Disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

1. The participant has a body weight within the 5th through 95th percentile by age, inclusive, as determined by the National Center for Health Statistics.
2. The participant must have a diagnosis of GERD prior to randomization and medical history of signs or symptoms of GERD for at least 3 months prior to screening, based on physical examination, current symptoms (eg, heartburn), or diagnostic tests (eg, pH or endoscopy). Notes in the medical records and/or other source documents, such as prior endoscopies, can be used to support the diagnosis and will be recorded in the electronic case report form (eCRF).
3. The participant has at least one moderate GERD symptom based on the GERD Symptom Assessment Investigator scale performed at screening.
4. The participant must be able to swallow study drug tablet with water.
5. Parent or legal guardian (ie, legally authorized representative [LAR]) is willing and able to complete the informed consent process and participants are able to comply with study procedures and visit schedule.
6. Female participants who have experienced menarche must have a negative pregnancy test and will be counseled on pregnancy avoidance.

Exclusion Criteria:

1. The participant has used prescription or non-prescription proton pump inhibitors (PPIs) or histamine-2 receptor antagonist (H2RAs) within 7 days prior to randomization or requires use during the Treatment Period.
2. The participant has used sucralfate, or antacids within 1 day prior to randomization or requires their use during the Treatment Period.
3. The participant has received other agents affecting digestive organs, including muscarinic antagonists (eg, hyoscyamine), prokinetics, oral anticholinergic agents, prostaglandins, bismuth from 30 days prior to Day 1 or requires their use during the course of the study.
4. The participant has received atazanavir sulfate or rilpivirine hydrochloride from 5 days prior to Day 1 or requires their use during the course of the study.
5. The participant has received any investigational compound (including vonoprazan) within 30 days prior to the start of the Screening Period.
6. The participant is an immediate family member or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, child, sibling) or participant may have consented under duress.
7. The participant requires hospitalization or has surgery scheduled during the course of the study or has undergone major surgical procedures within 30 days prior to the Screening Period.
8. The participant has undergone prior gastrointestinal surgeries.
9. The participant has any abnormal laboratory test values that are considered clinically significant in the opinion of the investigator during the Screening Period.
10. The participant has a history of hypersensitivity or allergies to vonoprazan (including the formulation excipients: D-mannitol, microcrystalline cellulose, hydroxypropylcellulose, fumaric acid, ascorbic acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 8000, and titanium dioxide, or red or yellow ferric oxide).
11. The participant has used any prescription or over-the-counter medications (including herbal or nutritional supplements), other than those already excluded in criteria 1 to 5 above, within 14 days before the first dose of study drug or throughout the study. That is, unless the medication(s) is permitted by the sponsor following a review of available data which confirms concomitant administration of the medication is unlikely to affect either the safety of the participant or the pharmacokinetics of vonoprazan.
12. The participant has consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or other food products that may be CYP3A4 inhibitors (eg, vegetables from the mustard green family [kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 7 days (or 5 half-lives) before the first dose of study drug or throughout the study.
13. The participant has positive results at screening for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus (HCV).
14. The participant has severe renal impairment (estimated glomerular filtration rate < 30 mL/min).
15. The participant has moderate to severe hepatic impairment (Child-Pugh Class B and Child-Pugh Class C).
16. The participant has any of the following abnormal laboratory test values at the start of the Screening Period:

    1. Creatinine levels: >0.8 mg/dL (>70 μmol/L).
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) or total bilirubin >2 × ULN (except participants with Gilbert Syndrome).
17. In the opinion of the investigator, the participant is not suitable for entry into the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Strada Patient Care Center, Mobile, Alabama
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Med Research Associates, Inc, Hollywood, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - International Center for Research, Tampa, Florida
  - Children's Center for Digestive Health Care, LLC, Atlanta, Georgia
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Advantage Clinical Trials, The Bronx, New York
  - PriMED Clinical Research, Dayton, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Maspons Pediatric Gastro, El Paso, Texas
  - Stryde Research - NxT Step Pediatrics, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 22 participants were enrolled at 6 study sites in the United States between November 2023 and April 2024.
Groups:
- Vonoprazan 10 mg: Participants received vonoprazan 10 mg once daily (QD) for 14 days.
- Vonoprazan 20 mg: Participants received vonoprazan 20 mg QD for 14 days.
Period: Overall Study
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg
Started | 11 | 11
Completed | 10 | 9
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Voluntary Withdrawal | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set: includes all participants who received at least 1 dose of study drug.
Groups:
- Vonoprazan 10 mg: Participants received vonoprazan 10 mg QD for 14 days.
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.92) | 8.6 (1.69) | 8.9 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 10 | 20
  Black or African American | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration at Steady-state (Cmax,ss) of Vonoprazan
Description: Plasma pharmacokinetic (PK) parameters were estimated using a non-linear mixed effects model and were determined from the concentration-time data for all evaluable participants. Actual sampling times, rather than scheduled or nominal sampling times, were used in all computations using sampling time. Data presented based on collections on both Day 7 and Day 14.
Time Frame: Day 7: pre-dose, 0.5 to 1.5 hour and 2.5 to 3.5 hours post dose; Day 14: pre-dose, 1 to 2 hours and 3 to 4 hours post dose
Population: PK Set: includes all participants who received at least 1 dose of study drug and had sufficient concentration data to support accurate estimation of at least 1 PK parameter.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg
Number analyzed (Participants) | 10 | 11
ng/mL | 16.2 [9.31 to 27.1] | 42.1 [10.1 to 72.7]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve During the Dosing Interval τ at Steady State (AUCτ,ss) of Vonoprazan
Description: Plasma PK parameters were estimated using a non-linear mixed effects model and were determined from the concentration-time data for all evaluable participants. Actual sampling times, rather than scheduled or nominal sampling times, were used in all computations using sampling time. Data presented based on collections on both Day 7 and Day 14.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg
Number analyzed (Participants) | 10 | 11
h*ng/mL | 88.3 [51.7 to 121] | 251 [72.1 to 549]

3. Primary Outcome: Apparent Oral Clearance (CL/F) at Steady State of Vonoprazan
Description: Oral PK parameters were estimated using a non-linear mixed effects model and were determined from the concentration-time data for all evaluable participants. Actual sampling times, rather than scheduled or nominal sampling times, were used in all computations using sampling time. Data presented based on collections on both Day 7 and Day 14.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: L/h
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg
Number analyzed (Participants) | 10 | 11
L/h | 125 [82.9 to 193] | 118 [36.4 to 278]

4. Primary Outcome: Apparent Central Volume of Distribution (Vz/F) at Steady State of Vonoprazan
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: liters
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg
Number analyzed (Participants) | 10 | 11
liters | 491 [227 to 828] | 444 [164 to 1310]

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: Safety Set: includes all participants who received at least 1 dose of study drug.
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vonoprazan 10 mg (N=11) | Vonoprazan 20 mg (N=11)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators (PIs) are not permitted to publish the data. Data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the PIs to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority over all such issues.

DOCUMENTS (2):
  • Study Protocol (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT06106022/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT06106022/SAP_001.pdf